CLINICAL TRIAL: NCT06416540
Title: The Effect of Upper Extremity Theraband Exercises on Respiratory Functions, Muscle Strength, Functional Mobility and Quality of Life in Intensive Care Patients
Brief Title: Upper Extremity Theraband Exercises in Intensive Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Betül Taşpınar, Study Director, Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICU-THERABAND-35
Record Dates: First submitted 2024-04-26; First posted 2024-05-16 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Exercise; Intensive Care Unit Patients
Keywords: Intensive Care Units; Exercise; Quality of Life; Physical Therapy Techniques
MeSH Terms: conditions — Motor Activity | interventions — Rehabilitation; Intensive Care Units; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theraband Exercises plus Conventional Physiotherapy and Rehabilitation Group (TB+CPRG) (Experimental): Upper Extremity Theraband Exercises Program Exercise training will be applied in a total of 3 sets, 30-60 min/session, 5 days/week, 8-10 repetitions/set, depending on the condition of each patient, during the patients' stay in the intensive care unit.
  Conventional Physiotherapy and Rehabilitation Program Normal joint range movements, airway clearing techniques, breathing exercises and mobilization will be applied to both groups included in the study by the physiotherapist. These movements will be performed once a day for 10 repetitions.
  Interventions: Other: Theraband Exercises plus Conventional Physiotherapy and Rehabilitation Program; Other: Conventional Physiotherapy and Rehabilitation Program
- Conventional Physiotherapy and Rehabilitation Group (CPRG) (Other): The control group will receive only conventional rehabilitation treatment. Although the duration of the session varies depending on the patient's condition, it will last approximately 30-60 minutes.
  Conventional Physiotherapy and Rehabilitation Program Normal joint range movements, airway clearing techniques, breathing exercises and mobilization will be applied to both groups included in the study by the physiotherapist. These movements will be performed once a day for 10 repetitions.
  Interventions: Other: Conventional Physiotherapy and Rehabilitation Program

INTERVENTIONS:
Other: Theraband Exercises plus Conventional Physiotherapy and Rehabilitation Program — Upper extremity, shoulder flexion, abduction, elbow flexion and wrist extension movements will be applied to the study group by the physiotherapist in combination with the breathing pattern. The program will start with yellow therabant and the difficulty level will be increased according to the patient's condition. Exercise training will be applied in a total of 3 sets, 30-60 min/session, 5 days/week, 8-10 repetitions/set, depending on the condition of each patient, during the patients' stay in the intensive care unit.
  Conventional Physiotherapy and Rehabilitation Program Normal joint range movements, airway clearing techniques, breathing exercises and mobilization will be applied to both groups included in the study by the physiotherapist. Hemodynamic and respiratory values for each level are monitored on the monitor. In addition, the patient will be monitored for symptoms such as blackness and dizziness by asking the patient.
  Other Names: Theraband Exercises in ICU
  Arms: Theraband Exercises plus Conventional Physiotherapy and Rehabilitation Group (TB+CPRG)
Other: Conventional Physiotherapy and Rehabilitation Program — Normal joint range movements, airway clearing techniques, breathing exercises and mobilization will be applied to both groups included in the study by the physiotherapist. Hemodynamic and respiratory values for each level are monitored on the monitor. In addition, the patient will be monitored for symptoms such as blackness and dizziness by asking the patient.
  Other Names: Control Group

SUMMARY:
Intensive Care Unit (ICU) is a special unit that deals with the diagnosis, treatment, and follow-up of patients who are in critical or severe condition and can not maintain their body balance. In this unit, appropriate examinations and treatments are applied to patients by experts using continuous monitoring and advanced technology 24 hours a day, 7 days a week. Immobilization is often a part of treatment in intensive care units. Long-term immobilization can lead to respiratory system problems such as mucociliary dysfunction, compromise of airway integrity, decreased lung capacity and decreased cough efficiency. Theraband exercises have been used in many settings as part of the therapeutic treatment of patients with poor motor abilities. However, there is not enough evidence in the literature as there is no study on the effectiveness of theraband exercises in the intensive care unit. Therefore, the aim of our study is; To examine the effects of upper extremity theraband exercises on respiratory functions, muscle strength, functional mobility and quality of life in intensive care patients.

DETAILED DESCRIPTION:
Intensive Care Unit (ICU) is a special unit that deals with the diagnosis, treatment and follow-up of patients who are in critical or severe condition and can not maintain their body balance. In this unit, appropriate examinations and treatments are applied to patients by experts using continuous monitoring and advanced technology 24 hours a day, 7 days a week. Patients who require constant cardiovascular monitoring, need mechanical ventilation and renal support, have major metabolic disorders, have head trauma, chest injuries or other multiple injuries are generally admitted to this unit. Although care in the intensive care unit reduces the mortality risk of patients by up to 60%, controlled mechanical ventilation can cause musculoskeletal problems due to reasons such as inactivity, sepsis, malnutrition, insulin resistance and systemic inflammation. Immobilization is often a part of treatment in intensive care units. Long-term immobilization can lead to respiratory system problems such as mucociliary dysfunction, compromise of airway integrity, decreased lung capacity and decreased cough efficiency. These problems are associated with factors such as sedation practices, artificial airway use, and airway obstruction. These factors disrupt natural airway clearing mechanisms, make it difficult to expel phlegm, and cause secretion accumulation. Accumulation of secretion may cause obstruction of the airways, increased respiratory resistance, alveolar hypoventilation, obstruction atelectasis and the development of pneumonia. Airway closure can lead to problems associated with body weight, decrease functional residual capacity, result in consolidation, changes in endotracheal tube position, pneumonia, lobar atelectasis, collapse, acute respiratory distress syndrome (ARDS), weakness of respiratory muscles, and lung volume loss due to acute lung injury. Loss of strength in the respiratory muscles in patients connected to mechanical ventilation frequently triggers lung complications such as atelectasis, pneumothorax and pneumonia. Decrease in respiratory function, continued muscle weakness, long-term mechanical ventilation and muscle contractures may negatively affect patients' quality of life. Inadequate or incomplete treatment is associated with recurrent symptoms. In addition, immobilization may also trigger neuromuscular weakness due to disuse atrophy, decreased muscle strength, and functional impairment. This weakness can range from severe paralysis, with or without loss of deep tendon reflexes. Acquired muscle weakness involves a complex mechanism. Factors such as immobility, local and systemic inflammation affect this process. During bed rest, the use of skeletal muscles decreases, which affects the morphology, contractility and aerobic capacity of the muscles, causing atrophy and muscle weakness. The period with the greatest loss of strength is the first week of immobilization. It has been observed that the quality of life of patients hospitalized in the intensive care unit for a long time decreases and their dependency increases while performing daily life activities. This condition has been associated with decreased mobility of patients as a result of muscle weakness and immobilization. According to studies in the literature, it can generally take an average of 12 months for patients' functional levels to improve after discharge. These findings emphasize the importance of factors that may affect the quality of life and daily living activities of patients who stay in the intensive care unit for a long time. Physiotherapists working in intensive care units deal with the complications and problems associated with this type of immobilization. Early rehabilitation plays an important role in the management of these patients to create an appropriate physiotherapy program, increase mobilization levels, reduce intensive care unit and hospital stays, and improve functional ability. In the systematic review and meta-analysis by Anekwe et al., in which they examined the effects of early rehabilitation on preventing the development of muscle weakness in the intensive care unit, it was revealed that physiotherapy applications in the intensive care unit reduced the development of acquired muscle weakness in the intensive care unit by a rate ranging from 29% to 37% in the randomized population. Physiotherapy and rehabilitation practices in intensive care address the basic problems of patients while also taking into account accompanying problems. Among the objectives of these interventions are to increase mobility, prevent muscle weakness and conditioning loss, optimize function, enhance mobility, clear airway secretions, reduce the frequency of atelectasis and pneumonia, maintain or regain lung volume, reduce respiratory workload, increase oxygen transport, and improve ventilation-perfusion matching. These interventions also aim to decrease and prevent dependence on mechanical ventilation, reduce and correct complications associated with immobility, minimize morbidity, improve quality of life, increase survival, and minimize the need for post-intensive care rehabilitation. In intensive care, physiotherapy and rehabilitation interventions often require the use of different modalities in combination. In these patients, resistance muscle training can increase muscle mass and force production. In order for these exercises to be effective, it is recommended to perform 3 sets of 8-10 repetitions at an intensity between 50% and 70% of the maximum repetition, in accordance with the patient's tolerance. Equipment such as elastic bands and free weights can be used to perform in-bed exercises, but the use of these equipment should be carefully managed for the comfort and safety of the patient. These exercises facilitate weaning from mechanical ventilation and help the patient gain maximum functional capacity. Muscle exercises applied in the intensive care unit are aimed at achieving goals such as being able to perform basic daily living activities and walking 20-50 meters independently. Exercise of the lower and upper extremities is performed in intensive care patients to maintain joint mobility, as well as to improve soft tissue resistance, muscle strength and functions, and to reduce the risk of thromboembolism. Lower extremity exercise training programs can increase muscle strength and endurance in patients with peripheral muscle weakness, which may improve quality of life. Upper extremity exercises should be included in the program due to their participation in daily life activities and support for breathing. These exercises target the upper body and arm muscles, as well as the respiratory muscles. Especially in patients with severe airway obstruction, the diaphragm must be supported by accessory respiratory muscles because it cannot create sufficient inspiratory pressure. Unsupported arm exercises can reduce the support of these muscles for breathing and affect the breathing pattern. The upper extremity exercise program may include various activities such as arm ergometer, free weights and elastic bands, thus increasing upper extremity endurance and strength. Theraband is an elastic band designed to be used for a variety of purposes, introduced by the Akron Hygenic company in 1978. These bands are available in different colors and resistance levels, allowing users to tailor their workouts to their needs and skill level. Theraband exercises have been used in many settings as part of the therapeutic treatment of patients with poor motor abilities. These exercises provide activation of antagonist, stabilizer and accessory muscles. One of the most distinctive features that distinguish these bands from other resistance devices is their ability to work independently of gravity. The resistance of this flexible exercise band varies depending on how much the user stretches and is therefore based on tension level, not gravity. As you stretch the Therabands, their resistance increases, so users can achieve their desired level of difficulty. When using elastic bands, difficulty levels vary depending on the stretched measurements. Additionally, the colors of these bands also guide users on their resistance levels. Therabands come in eight different colors, and each color represents a specific level of difficulty. The color sequence progresses from easy to difficult, including tan, yellow, red, green, blue, black, gray and golden yellow. This color-coding system allows users to choose a resistance level that suits their needs and skill level, and also helps them keep track of their progress. Theraband exercises are an attractive option that can be preferred in the intensive care unit because it is a cheap and simple technique. However, the application of theraband exercises in critical illness situations such as Intensive Care Units has not yet been described in detail. In a case report, it was shown that upper extremity theraband exercises applied to a patient in the intensive care unit for 31 days provided significant improvements in the patient's movements. It was also stated that the patient's ability to maintain a sitting position on the edge of the bed improved from the 27th day. For this reason, theraband exercises are thought to be a suitable, safe and applicable method to maintain upper extremity motor activities and improve trunk control. However, there is not enough evidence in the literature as there is no study on the effectiveness of theraband exercises in the intensive care unit. Therefore, the aim of our study is; To examine the effects of upper extremity theraband exercises on respiratory functions, muscle strength, functional mobility and quality of life in intensive care patients.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Being conscious
* Being clinically stable
* Not dependent on mechanical ventilation
* Being deemed suitable for physiotherapy and rehabilitation practices by an intensive care specialist

Exclusion Criteria:

* Having psychiatric disorders and extreme agitation
* Having cooperation disorders
* Having the progressive neuromuscular disease
* Having any trauma to the chest wall
* Having any deformity of the thorax that will affect breathing
* Having diseases that require constant use of sedative or analgesic agents
* Being in shock stiuation
* Having cardiac and respiratory instability (FiO₂> 55%, PaO₂< 65 mmHg, respiratory rate >30 breaths/min, systolic blood pressure >200 mmHg or <80 mmHg, diastolic blood pressure >100 mmHg or <50 mmHg)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Assessment of Consciousness | At baseline and on average day 10
  The patients' consciousness will be evaluated with the Glasgow coma scale. Scores between 3 and 7 indicate severe coma, between 8 and 11 indicate moderate coma, between 12 and 14 indicate mild coma, and 15 points indicate that the patient is not in a coma.
Assessment of Comorbidity | At baseline and on average day 10
  The Charlson Comorbidity Index (CKI) will be used to evaluate the patients' accompanying problems. The total CKI score varies between 0-33. As the score increases, the degree of comorbidity also increases.
Assessment of Disease Severity | At baseline and on average day 10
  APACHE II score is a measure used to estimate the severity of the disease and the risk of mortality, taking into account the patient's clinical condition and age. This score is based on an initial 12-component score and is evaluated on a range from 0 to 71 points. As the total APACHE II score increases, the severity of the patient's condition also increases.
Assessment of Respiratory Functions | At baseline and on average day 10
  Forced expiratory volume in the first second (FEV1), forced vital capacity (FVC), and the ratio of forced expiratory volume in the first second to forced vital capacity (FEV1/FVC) with spirometry will be evaluated.
Assessment of Peripheral Muscle Strength | At baseline and on average day 10
  Upper and lower extremity peripheral muscle strength will be evaluated with the Medical Research Council (MRC) scale, which is a manual muscle testing method. Each muscle group is classified between 0 (complete paralysis) and 5 (normal muscle strength) points. The total MRC scale score is evaluated between 0 and 60. MRC score <48 points indicates muscle weakness.
Assessment of Functional Mobility | At baseline and on average day 10
  Mobilization status of the participants will be evaluated using the ICU Mobility Scale. The scale includes 11 different mobility levels. These levels range from passive mobilization (0: bedridden) to independent mobilization (10: active mobilization without assistance). As the YMS score increases, the mobility level also increases
Assessment of Quality of Life | At baseline and on average day 10
  Participants' quality of life will be assessed using the Nottingham Health Profile (NSP). NSP is a quality of-life scale that aims to evaluate a person's self-perceived health status in emotional, physical, and social aspects. The total score varies between 0-600, and higher scores indicate worse quality of life.
Assessment of Anxiety and Depression Status | At baseline and on average day 10
  The anxiety and depression status of the participants will be evaluated using the Hospital Depression and Anxiety Score (HADS). The scale has two subparameters: anxiety (HAD-A) and depression (HAD-D). It consists of fourteen items, seven of which investigate symptoms of depression and seven of which investigate symptoms of anxiety. Answers are scored between 0-3. 0-1 is considered healthy, 2 is borderline and 3-4 is considered sick. As a result of the studies, the cut-off score for the anxiety subscale was found to be 10, and the cut-off score for the depression subscale was found to be 7. Patients can score a minimum of '0' and a maximum of '21' from two subscales.
Assessment of respiratory muscle strength | At baseline and on average day 10
  Voluntary measurement of respiratory muscle strength will be made with a portable, electronic mouth pressure measurement device. Maximum static inspiratory pressure (MIP) and maximum static expiratory pressure (MEP) measurement are practical, voluntary measurement methods frequently used in the clinic to measure the strength of the inspiratory and expiratory muscles. The highest pressure value from the measurements will be selected for analysis.
Assessment of thoracic mobility | At baseline and on average day 10
  For thoracic mobility, the circumference of the thorax will be measured with a tape measure after expiration and inspiration.
Assessment of fatigue | At baseline and on average day 10
  Patients' general perception of body fatigue and dyspnea will be recorded with the Modified Borg scale. A value of 0 indicates no dyspnea and fatigue, and a value of 10 indicates severe dyspnea and fatigue.
Assessment of hand grip strength | At baseline and on average day 10
  The patients' hand grip strength will be measured with a Jamar hydraulic hand dynamometer. With the help of the device, measurements will made three times in both hands of the patient and the grip strength is determined by taking the average.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar Unde Ayvat, Assoc. Prof., Principal Investigator — Izmir Democracy University; Ferruh Taspinar, Prof. Dr., Principal Investigator — Izmir Democracy University
Locations (1):
- Betül TAŞPINAR, Konak, İ̇zmi̇r, Turkey (Türkiye)